CLINICAL TRIAL: NCT06101433
Title: The Effect of Soy Isoflavones on Non-alcoholic Fatty Liver Disease and the Level of Fibroblast Growth Factor-21 and Fetuin A
Brief Title: The Effect of Soy Isoflavones on Non-alcoholic Fatty Liver Disease and the Level of FGF-21 and Fetuin A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Asal Neshatbini Tehrani, Principal Investigator, Ahvaz Jundishapur University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATehrani
Record Dates: First submitted 2023-10-11; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: NAFLD
Keywords: Non-alcoholic fatty liver disease; Isoflavones; Soy foods; FGF21; Liver steatosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Soybean Proteins

STUDY DESIGN:
Intervention Model Description: Patients were randomly classified into placebo or soy isoflavone groups using block randomization stratified by menopause status and gender for 12 weeks
Who Masked: Participant, Investigator
Masking Description: The participants and investigator were blinded to study groups (double blinded study)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The placebo group (Placebo Comparator): Subjects in the placebo group, were advised to take two placebo tablets per day for 12 weeks along with life style modification such as physical activity of 30 minutes for 3 days per week with medium intensity and food intake consults provided by clinical guidelines of NIH and the North American Association for the Study of Obesity. The placebo tablets contained starch and they were similar to the soy isoflavone tablets in smell, taste, and appearance. The placebo tablets were made by Gol Daru Pharmaceutical Company, Isfahan, Iran.
  Interventions: Other: Placebo
- The soy isoflavone group (Active Comparator): In the soy isoflavone group, patients took 100 mg soy isoflavone in the form of two tablets per day for 12 weeks along with lifestyle modification. Each soy isoflavone 50 mg tablet contained 1.49 mg of genistein, 31.86 mg of genistin, 1.75 mg of daidzein, 13.21 mg of daidzin, 0.55 mg of glycitein and 1.14 mg of glycitin. The soy isoflavone tablets were made by Gol Daru Pharmaceutical Company, Isfahan, Iran.
  Interventions: Dietary Supplement: Soy isoflavone

INTERVENTIONS:
Dietary Supplement: Soy isoflavone — the subjects in the soy isoflavone group were told to take 2 drugs per day, one in the morning after the breakfast and one at night after the dinner and continue this pattern for 12 weeks.
  Other Names: Soyagol
  Arms: The soy isoflavone group
Other: Placebo — the subjects in the placebo group were told to take 2 placebo tablets per day, one in the morning after the breakfast and one at night after the dinner and continue this pattern for 12 weeks.
  Arms: The placebo group

SUMMARY:
In this research, the investigators tested the effect of 12-week supplementation with soy isoflavones on non alcoholic fatty liver disease (NAFLD) management and the level of fibroblast growth factor-21 (FGF-21) and fetuin A as markers of NAFLD progression.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) accounts as a crucial health concern with a huge burden on health and economic systems. The aim of the present study was to investigate the effect of soy isoflavone intake on hepatic outcomes and the level of fibroblast growth factor-21 (FGF-21) and fetuin A in patients with NAFLD. Fifty patients with NAFLD were randomized to either receive two tablets of soy isoflavone (100 mg/d) or placebo. Dietary intakes, anthropometric parameters, the serum levels of liver function tests including alanine amino transferase (ALT), aspartate amino transferase (AST) and gamma glutamyl transferase (GGT), FGF-21, fetuin A and hepatic histological features by Fibroscan assessed at study initiation and after week 12.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* without any history of allergy to soy or excessive consumption of soy products
* without chronic diseases including renal, liver, heart, respiratory, cardiovascular, malignancies, auto immune disorders, cushing's syndrome, thyroid dysfunction, hepatitis, cirrhosis, biliary disorders, diabetes, gastrointestinal tract diseases affecting the gut absorption and psychiatric disorders considering as an obstacle for patients to prepare written informed consent;
* hepatic steatosis grade 2 and higher with fibroscan confirmation (CAP > 260 dB/m);
* without history of excessive alcohol drink (≥10 g/day);
* without history of drug consumption with approved positive effects on NAFLD treatment (i.e. metformin, vitamin E, ursodeoxycholic acid, phenytoin, tamoxifen, lithium, corticosteroids and methotrexate) in last three months;
* without the history of bariatric surgery or following weight loss diets within 6 months;
* without history of smoking;
* not being a pregnant or lactating woman

Exclusion Criteria:

* consuming less than 90% of intended supplements.
* unwillingness for study collaboration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Hepatic histological features by Fibroscan | 12 weeks
  The subject's hepatic histological features using Fibroscan (Echosense, France) assessed at study initiation and at week 12.
The Level of serum liver enzymes | 12 weeks
  The serum levels of alanine amino transferase (ALT), aspartate amino transferase (AST) and gamma glutamyl transferase (GGT) measured through enzymatic methods by Delta Darman Part test kits (Delta darman part, Tehran, Iran) at study initiation and at the end of the trial

SECONDARY OUTCOMES:
fibroblast growth factor-21 (FGF-21) | 12 weeks
  The serum level of FGF-21 measured via ELISA commercial kits (ZellBio GmbH Veltlinerweg 29, 89075, Ulm, Germany) at study initiation and at week 12.
Fetuin A | 12 weeks
  The serum level of fetuin A measured via ELISA commercial kits (ZellBio GmbH Veltlinerweg 29, 89075, Ulm, Germany) at study initiation and at week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Asal Neshatbini Tehrani, PhD, Principal Investigator — Ahvaz Jundishapur University of Medical Sciences
Locations (1):
- Asal Neshatbini Tehrani, Ahvāz, Khuzestan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Raw data that support the findings of this study are available from the corresponding author, upon reasonable request by contacting the principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Raw data that support the findings of this study are now available from the principal investigator
Access Criteria: upon reasonable request by contacting the principal investigator